CLINICAL TRIAL: NCT07264400
Title: Impact of Physical Activity During Pregnancy on Cardiac Variability in Newborns
Acronym: NEOMOUV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2025 PAYSAL; 2025-A00329-40 (Other: ANSM)
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Newborn Infant
Keywords: heart rate variability; oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of cardiorespiratory function (Experimental): A Holter ECG and oximetry recording will be performed on the child's second night for a minimum of 6 hours. Three electrodes will be placed on the newborn's chest, along with a pulse oximeter, and removed the following day.
  Parents will be contacted by email at the child's second birthday to obtain information on their child's height and weight growth, and their neurodevelopment will be assessed using the Age and Stage Questionnaire (ASQ-3) at 24 months.
  Interventions: Other: Heart rate variability; Other: Pulmonary function

INTERVENTIONS:
Other: Heart rate variability — A Holter ECG recording will be performed on the child's second night for a minimum of 6 hours.
Other: Pulmonary function — Oximetry recording will be performed on the child's second night for a minimum of 6 hours.

SUMMARY:
Ancillary study of the PregMouv study which aims to evaluate an intervention allowing the best adherence of women in terms of physical activity. Several types of interventions are therefore planned in this study: no intervention, physical activity sessions in person, by videoconference or mixed (in person and videoconference) with accelerometer assessment of the level of physical activity practiced (in the form of energy expenditure, in MET). Thus, for our ancillary study, a comparison of the cardiac variability of newborns will be carried out according to the level of physical activity practiced by the mother regardless of the intervention she benefited from within the framework of the PregMouv study. A comparison of the average saturation and the time spent below 90% saturation will be carried out via a continuous recording of saturation by oximetry. A longitudinal follow-up for the assessment of height and weight growth (from growth curves) and neurodevelopment (by clinical examination and self-questionnaire) is also planned until the child is 2 years old.

DETAILED DESCRIPTION:
Holter ECG and oximetry recording of the newborn for a minimum of 6 hours during their stay in the maternity ward, or in another perinatal sector. Evaluation at the child's 2nd birthday by collecting the height-weight curve, the 2nd birthday clinical examination and self-questionnaire, ASQ, from the parents. Blind interpretation and analysis of the results. Comparison of the results according to the mothers' level of physical activity (in MET/min/week), assessed by the accelerometer study at T2 and T3 of pregnancy. Search for correlation between the level of physical activity practiced and the child's physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* All newborns of mothers who participated in the PregMouv study and who have at least one piece of data for the main criterion from the PregMouv study (physical activity at T1/T2),
* born at the Clermont Ferrand University Hospital and after parental agreement for their child to participate may be included.

Exclusion Criteria:

* Newborns requiring aminergic support in the first days of life,
* making heart rate variability analysis impossible,
* having received invasive ventilatory support that does not allow analysis of the oximetry recording.
* Parental refusal or inability of parents to give their consent for their child to participate.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | during the child's second night.
  Is measured by SDNN (standard deviation of all normal R-R intervals), a reflection of the variability of the global autonomic nervous system of newborns, obtained from a Holter ECG recording.

SECONDARY OUTCOMES:
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by RMSSD (root mean square of differences of successive RR intervals)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by NN50 (number of RR intervals that differ by > 50 ms)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by p NN50 (percentage of consecutive RR intervals that differ by >50 ms)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by SD1 (standard deviation 1)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by and HF (high frequency power)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by SD2 (standard deviation 2)
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by SD1/SD2 ratio
Heart rate variability | during the child's second night
  Others parameters of heart rate variabilt obtained from a Holter ECG recording by LF (low frequency)
Respiratory function | During the child's second night
  Assessed by oximetry: desaturation index and drop per hour of more than 3%.
Respiratory function | During the child's second night
  Assessed by oximetry: time spent below 90%, 80% and 70% saturation (in raw value and in two classes depending on whether the value is greater than or equal to 5)
Respiratory function | During the child's second night
  Assessed by oximetry: mean saturation (in raw value and in two classes depending on whether the value is strictly less than 93)
Height growth | at 2 years old
  height measurement in centimeters
weight growth | at 2 years old
  weight measurement in kilograms
neurodevelopment | at 24 months
  assessed by the Ages & Stages Questionnaires, Third Edition (ASQ-3)

CONTACTS AND LOCATIONS:
Overall Officials: Justine Paysal, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No